CLINICAL TRIAL: NCT01459718
Title: A Multicenter Open Label Phase II Study to Evaluate the Safety and Efficacy of Deferasirox in Combination With Deferoxamine Followed by Transitioning to Deferasirox Monotherapy in β-thalassemia Patients With Severe Cardiac Iron Overload
Brief Title: Safety and Efficacy of Deferasirox in Combination With Desferoxamine in β-thalassaemia Patients With Severe Cardiac Iron Overload
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study terminated due to low enrollment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AGR02; 2009-018091-34 (EudraCT Number)
Record Dates: First submitted 2011-07-20; First posted 2011-10-26 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Transfusion-dependent β-thalassemia Patients; Cardiac Iron Overload
Keywords: Severe cardiac iron overload; deferasirox; β-thalassaemia; cardiac dysfunction
MeSH Terms: interventions — Deferasirox; Deferoxamine

ARMS (1):
- Deferasirox / Deferasirox + Deferoxamine (DFO) (Experimental): During Phase A, the induction treatment at entry, participants received Deferasirox -DFO combination. During Phase B, when participants transitioned to less intensive chelation therapy, participants received Deferasirox monotherapy.
  Interventions: Drug: Deferasirox; Drug: Deferoxamine (DFO)

INTERVENTIONS:
Drug: Deferasirox — 20-40 mg/kg/day orally, once daily
  Other Names: ICL670, Exjade
Drug: Deferoxamine (DFO) — 40 mg/kg/day subcutaneous (sc) infusion, 3-4 days per week
  Other Names: DFO, Desferal

SUMMARY:
The primary efficacy endpoint of this interventional study was to evaluate the number of patients achieving a complete response (CR), defined as patients switching from intensive deferasirox -DFO treatment, at any time point during the 24 months of study, to deferasirox monotherapy based on improvement in the cardiac magnetic resonance imaging (MRI) T2* value to >10ms, and continue to maintain their MRI T2* to values >10 msec.

DETAILED DESCRIPTION:
This study was planned to recruit 52 transfusion-dependent β-thalassemia patients with severe cardiac iron overload. However only 13 patients participated in the study during a 3 year and 5 month timeframe. The study was terminated due to the slow enrollment rate due to scarcity of the patient population with severe cardiac iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with β-thalassemia major, at least 18 years old, having given written consent to participate in the study.
* Cardiac MRI T2* value ranging from <=4 to <=10 ms.
* LVEF ≥ 56 % as determined by CMR.
* Patients with LIC > 10mg Fe/g dw will be included in the protocol. Study will evaluate the first 10 patients at 6 months, and if no safety signals are present, patients with LIC>5 mg Fe/g dw will be allowed to be included.
* Prior iron chelation treatment with DFO, DFP, DFX or combination DFO-DFP

Exclusion Criteria:

* Patients with symptoms of cardiac dysfunction symptoms (shortness of breath at rest or exertion, orthopnea, exercise intolerance, lower extremity edema, arrhythmias).
* Patients with cardiac T2* MRI < 4 or > 10 ms.
* Patients not compliant to intensive iron chelation therapy regimens such i.v DFO 24 hr infusions or DFO-DFP combination.
* Patients with documented liver failure (presence of portal hypertension, hepatic edemas, ascites).
* Patients unable to undergo study assessments, including blood sampling, MRI, e.g., are claustrophobic to MRI, have a pacemaker, ferromagnetic metal implants other than those approved as safe for use in MRI scanners (e.g., some types of aneurysm clips, shrapnel in proximity to vital organs such as the retina), are obese (exceeding the equipment limits).
* Patients with serum creatinine > ULN or with significant proteinuria as indicated by a urinary protein/creatinine ratio ≥ 1.0 in a non-first void urine sample at baseline. Patients with creatinine clearance <60 ml/min will be excluded.
* Patients with ALT (SGPT) levels > 5 x ULN.
* Patients with considerable impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral deferasirox / ICL670 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection.
* History or clinical evidence of pancreatic injury or pancreatitis.
* Patients with a known hypersensitivity to any of the study drugs or the drug's excipients.
* History of clinically relevant ocular and/or auditor toxicity related to iron chelation therapy.
* Patients with psychiatric or addictive disorders which prevent them from giving their informed consent or undergoing any of the treatment options or patients unwilling or unable to comply with the protocol.
* Patients with a known history of HIV seropositivity (Elisa or Western blot).
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Female patients who are pregnant or breast feeding.
* Female patients of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test ≤ 48 hours prior to the study drugs.
* Patients participating in another clinical trial or receiving an investigational drug.
* History of non-compliance with medical regimens or patients who are considered potentially unreliable and/or not cooperative, unwilling or unable to comply with the protocol.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this open-label, single arm study 31 participants were enrolled (one participant was screened twice and was assigned 2 screening numbers; therefore the number enrolled = 32). Of these enrolled participants, 13 were randomized.
Period: Overall Study
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Started | 13
Safety Analysis Set | 13
Completed | 10
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving a Complete Response (CR)
Description: Complete Response is defined as patients that stop intensive deferasirox -DFO treatment, at any time point during the 24 months of study, based on an improvement in the cardiac Magnetic Resonance Imaging T2 star technique (MRI T2*) value being >10ms, and continue to be treated with deferasirox monotherapy without any further need for reverting back to intensive iron chelation treatment during the 24 months of study.
Time Frame: 24 months
Population: The full analysis set included all the participants entered in the study with at least a valid post-baseline assessment of the primary efficacy variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
Participants | 4

2. Primary Outcome: Number of Patients Achieving a Partial Response (PR)
Description: Partial Response is defined as patients that stop intensive deferasirox -DFO treatment at any time point during the 24 months study and transition to receive deferasirox monotherapy, but due to a deterioration in cardiac MRI T2* to a value < 10 ms revert back to intensive deferasirox -DFO iron chelation therapy during the 24 months of study.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
Participants | 0

3. Primary Outcome: Number of Patients With Stable Disease (SD)
Description: Stable Disease is defined as those patients that never achieved an improvement in the cardiac MRI T2* to values >10ms during the 24 months of study.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
Participants | 8

4. Secondary Outcome: Change From Baseline in Cardiac Iron Overload of Patients in Intensive Iron Chelation Therapy Consisting of Deferasirox-DFO and After Transition to Deferasirox Monotherapy
Description: Cardiac iron overload was determined by cardiac MRI T2*. Cardiac iron overload also was measured by the monthly velocity of heart MRI T2*.
Time Frame: Baseline, 6, 12, 18, 24 months
Population: The full analysis set included all the participants entered in the study with at least a valid post-baseline assessment of the primary efficacy variable. Here 'n' number analyzed signifies number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
Milliseconds (ms)
  6 months | 0.1 (1.4)
  12 months: number analyzed (Participants) | 10
  12 months | 0.7 (1.9)
  18 months: number analyzed (Participants) | 11
  18 months | 1.3 (2.4)
  24 months: number analyzed (Participants) | 10
  24 months | 2.4 (3.9)

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from baseline when the participant had severe cardiac iron overload to the time when the participant achieved mild/moderate cardiac overload (T2*>10 milliseconds [ms]).
Time Frame: 24 months
Population: The full analysis set included all participants entered in the study with at least a valid post-baseline assessment of the primary efficacy variable. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure at the specified time-point.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 5
ms | 13.0 (1.1)

6. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC)
Description: Change from baseline in LIC was determined by change in liver MRI T2*.
Time Frame: Baseline, 6, 12, 18, 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg of iron/gram of dry weight of liver
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
mg of iron/gram of dry weight of liver
  6 months | -5 (7.7)
  12 months: number analyzed (Participants) | 10
  12 months | -10.3 (9.2)
  18 months: number analyzed (Participants) | 11
  18 months | -10.2 (10.7)
  24 months: number analyzed (Participants) | 10
  24 months | -12.4 (10.1)

7. Secondary Outcome: Correlation Between Change From Baseline in Serum Ferritin and LIC Levels
Description: Spearman correlation coefficients between serum ferritin and LIC changes from baseline levels were reported.
Time Frame: Baseline, 6, 12, 18, 24 months
Population: Full analysis set included all participants entered in study with at least a valid post-baseline assessment of the primary efficacy variable. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable at each time point.
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 11
Spearman correlation coefficient
  6 months | 0.091
  12 months: number analyzed (Participants) | 9
  12 months | -0.033
  18 months | 0.347
  24 months: number analyzed (Participants) | 10
  24 months | 0.273

8. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF % was measured by cardiac magnetic resonance (CMR).
Time Frame: 6, 12, 18, 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of ejection fraction
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Number analyzed (Participants) | 12
Percentage of ejection fraction
  Baseline | 65 (4.4)
  6 months | 65.4 (5)
  12 months: number analyzed (Participants) | 10
  12 months | 64.8 (4.6)
  18 months: number analyzed (Participants) | 11
  18 months | 65.1 (4.8)
  24 months: number analyzed (Participants) | 10
  24 months | 66.2 (4.6)

ADVERSE EVENTS:
Arm/Group | Deferasirox / Deferasirox + Deferoxamine (DFO)
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox / Deferasirox + Deferoxamine (DFO) (N=13)
Haemolysis (Blood and lymphatic system disorders) | 1
Cardiac discomfort (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lithotripsy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox / Deferasirox + Deferoxamine (DFO) (N=13)
Thrombocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 6
Gastric disorder (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Discomfort (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 4
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Viral infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1
Muscle contusion (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Facial neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hypotonia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Genital burning sensation (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 2
Tooth repair (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
Study was terminated. Efficacy was not powered for analysis due to the low enrollment of only 13 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.